CLINICAL TRIAL: NCT01644565
Title: A Phase 1 Dose Escalating Study of Two Enterotoxigenic Escherichia Coli Prototype Adhesin-based Vaccines With or Without Modified Heat-labile Enterotoxin by Intradermal or Transcutaneous Immunization
Brief Title: Safety Study of Chimeric Vaccine to Prevent ETEC Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-12-07; S-12-07 (Other: Sponsor); NMRC.2012.0005 (Other: Naval Medical Research Center Institutional Review Board); 1924 (Other: Walter Reed Army Institute of Research Institutional Review Board)
Record Dates: First submitted 2012-07-11; First posted 2012-07-19 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Escherichia Coli Infection
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Group A-1 (Experimental): Recombinant fimbrial adhesin dscCfaE: 1 ug of dscCfaE ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE
- Group A-2 (Experimental): Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5: 2.6 ug of Chimera ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5
- Group A-3 (Experimental): Modified E. coli heat labile enterotoxin LTR192G: 100 ng of LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group B-1 (Experimental): Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 1 ug of dscCfaE + 100 ng of LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group B-2 (Experimental): Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5 and Modified E. coli heat labile enterotoxin LTR192G: 2.6 ug of Chimera + 100 ng of LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group C-1 (Experimental): Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 5 ug of dscCfaE + 100 ng of LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group C-2 (Experimental): Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5 and Modified E. coli heat labile enterotoxin LTR192G: 12.9 ug of Chimera + 100 ng of LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group D-1 (Experimental): Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 25 ug dscCfaE + 100 ng LTR192G ID on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group D-2 (Experimental): Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 1250 ug dscCfaE + 50 ng LTR192G TCI on study days 0, 21 and 42
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G

INTERVENTIONS:
Biological: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5
  Other Names: Chimera
  Arms: Group A-2; Group B-2; Group C-2
Biological: Recombinant fimbrial adhesin dscCfaE
  Other Names: dscCfaE
  Arms: Group A-1; Group B-1; Group C-1; Group D-1; Group D-2
Biological: Modified E. coli heat labile enterotoxin LTR192G
  Other Names: LTR192G
  Arms: Group A-3; Group B-1; Group B-2; Group C-1; Group C-2; Group D-1; Group D-2

SUMMARY:
The purpose of the study is to determine if immunization with a chimeric E. coli protein, dsc14CfaE-sCT2/LTB5, is safe and immunogenic when administered by vaccination under the skin.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and immunogenicity of dsc14cfaEsCTA2/LTB5 (Chimera) and dscCfaE administered with and without LTR192G by intradermal (ID) immunization and to gather additional data on the administration of dsCfaE and LTR192G via transcutaneous immunization (TCI) route. If vaccines are found to be safe and adequately immunogenic in humans, a down-selection would occur and a phase 2b vaccination/challenge study would be undertaken to further evaluate vaccine safety and allow a preliminary assessment of efficacy of one of these candidates by the ID or TCI route. With favorable evidence for safety, immunogenicity, efficacy, complemented by advances in standard methodology to combine multiple adhesins with an appropriate LT enterotoxoid form, a multivalent vaccine would be constructed and evaluated for further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved > 70% accuracy).
* Signed informed consent document.
* Available for the required follow-up period and scheduled clinic visits.
* Women: Negative pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within three (3) months following study completion.

Exclusion Criteria:

* Health problems (for example, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension or any other conditions that might place the subjects at increased risk of adverse events. Study clinicians, in consultation with the PI, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the Research Monitor as appropriate.
* Clinically significant abnormalities on physical examination.
* Use of immunosuppressive medications (systemic corticosteroids or chemotherapeutics that may influence antibody development), or immunosuppressive illness, including IgA deficiency (defined by serum IgA below the detectable limit).
* Women who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last study safety visit and currently nursing women.
* Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) 30 days before planned date of first vaccination or anytime through the last study safety visit.
* Positive blood test for HBsAg, HCV, HIV-1.
* Clinically significant abnormalities on basic laboratory screening.
* Exclusionary skin history/findings that would confound assessment or prevent appropriate local monitoring of AEs, or possibly increase the risk of an AE.
* History of chronic skin disease (clinician judgment).
* History of atopy such as active eczema.
* Acute skin infection/eruptions on the upper arms including fungal infections, severe acne or active contact dermatitis.
* Allergies that may increase the risk of AEs.
* Regular use (weekly or more often) of antidiarrheal, anti-constipation, or antacid therapy.
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* Prior exposure to ETEC or Vibrio cholera.
* History of microbiologically confirmed ETEC or cholera infection.
* Travel to countries where ETEC or V. cholera or other enteric infections are endemic (most of the developing world) within two years prior to dosing clinician judgment).
* Received previous experimental ETEC or V. cholera vaccine or live ETEC or V. cholera challenge.
* Occupation involving handling of ETEC or V. cholera currently, or in the past 3 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro L. Gutierrez, MD, MPH, Principal Investigator — Enteric Diseases Department, Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research Clinical trial Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 subjects were enrolled. An additional 2 subjects per cohort for Cohorts A-C and 2 subjects per group in Cohort D were included as alternates.
Groups:
- Group A-1: Recombinant fimbrial adhesin dscCfaE: 1 ug of dscCfaE ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dscCfaE
- Group A-2: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5: 2.6 ug of Chimera ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5
- Group A-3: Modified E. coli heat labile enterotoxin LTR192G: 100 ng of LTR192G ID on study days 0, 21 and 42
  Modified E. coli heat labile enterotoxin LTR192G
- Group B-1: Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 1 ug of dscCfaE + 100 ng of LTR192G ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dscCfaE
  Modified E. coli heat labile enterotoxin LTR192G
- Group B-2: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5 and Modified E. coli heat labile enterotoxin LTR192G: 2.6 ug of Chimera + 100 ng of LTR192G ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5
  Modified E. coli heat labile enterotoxin LTR192G
- Group C-1: Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 5 ug of dscCfaE + 100 ng of LTR192G ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dscCfaE
  Modified E. coli heat labile enterotoxin LTR192G
- Group C-2: Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5 and Modified E. coli heat labile enterotoxin LTR192G: 12.9 ug of Chimera + 100 ng of LTR192G ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dsc14CfaE-sCTA2/LTB5
  Modified E. coli heat labile enterotoxin LTR192G
- Group D-1: Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: 25 ug dscCfaE + 100 ng LTR192G ID on study days 0, 21 and 42
  Recombinant fimbrial adhesin dscCfaE
  Modified E. coli heat labile enterotoxin LTR192G
- Group D-2: Recombinant fimbrial adhesin dscCfaE and Modified E. coli heat labile enterotoxin LTR192G: TBD ug dscCfaE + 50 ng LTR192G TCI on study days 0, 21 and 42
  Recombinant fimbrial adhesin dscCfaE
  Modified E. coli heat labile enterotoxin LTR192G
Period: Overall Study
Arm/Group | Group A-1 | Group A-2 | Group A-3 | Group B-1 | Group B-2 | Group C-1 | Group C-2 | Group D-1 | Group D-2
Started | 5 | 5 | 5 | 5 | 5 | 7 | 7 | 10 | 8
Completed | 4 | 5 | 5 | 4 | 4 | 7 | 7 | 8 | 7
Not Completed | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Not completed — Undisclosed Medical History | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Family emergency | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Relocation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics within Final Clinical Study Report were not broken out by groups or cohorts. No randomization was presented to detail which subject was in which group or cohort. Data is presented as it was detailed in the FCSR. No explanation was given as to why groups were combined to report demographic data.
Groups:
- All Study Cohorts: Baseline data within Final Clinical Study Report was not broken out by groups or cohorts. No randomization was presented to detail which subject was in which group or cohort. Data is presented as it was detailed in the FCSR.
Arm/Group | All Study Cohorts
Number analyzed (Participants) | 57
Age, Customized [Number; unit: participants]
  Age 18 - 45 years | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 30
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Safety - Occurrence of Adverse Events
Description: Occurrence of related and unrelated to vaccine AE's
Time Frame: 1 year
Measure: Number; unit: Number of Adverse Events
Arm/Group | Group A-1 | Group A-2 | Group A-3 | Group B-1 | Group B-2 | Group C-1 | Group C-2 | Group D-1 | Group D-2
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 4 | 7 | 7 | 8 | 7
Number of Adverse Events
  Related to Vaccine | 7 | 21 | 19 | 20 | 18 | 23 | 25 | 38 | 25
  Unrelated to Vaccine | 17 | 14 | 16 | 14 | 10 | 20 | 8 | 20 | 26

2. Secondary Outcome: Number of Participants With Immune Responses to Vaccine Antigens
Description: Number of participants with immune responses to vaccine antigens from baseline. Peripheral blood mononuclear cells (PBMCs) were collected to determine IgA antibody secreting cells (ASC) responses to dscCfaE and LTB. For each antigen, pre-and post-dosing samples were tested for total and vaccine-specific numbers of IgA-ASCs using the ELISPOT assay. A positive IgA-ASC response was defined as a > 2-fold increase over the baseline value of the ASC per 10^6 PBMC, when the number of ASC was >0.5 per 10^6 in the baseline sample. When the number of baseline ASCs was less than 0.5 per 10 PBMC, a subject was considered a responder if the post-vaccination value was greater than 1.0 per 10^6 PBMC.
Time Frame: baseline and post dose
Population: A total of 55 subjects across cohorts received the minimum required 2 doses of investigation product(s) and were evaluable for the immunology analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A-1 | Group A-2 | Group A-3 | Group B-1 | Group B-2 | Group C-1 | Group C-2 | Group D-1 | Group D-2
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 7 | 7 | 10 | 7
Participants
  Serum IgG (aCfaE) - >4-fold rise in baseline titer | 0 | 5 | 0 | 4 | 4 | 7 | 7 | 9 | 7
  Serum IgG (aLT) - >4-fold rise in baseline titer | 0 | 5 | 5 | 5 | 4 | 7 | 7 | 9 | 3
  Serum IgA (aCfaE) - >4-fold rise in baseline titer | 0 | 1 | 0 | 3 | 2 | 3 | 3 | 5 | 0
  Serum IgA (aLT) - >4-fold risein baseline titer | 0 | 3 | 3 | 4 | 4 | 5 | 7 | 7 | 6
  IgA ASC (aCfaE) - >2-fold increase over baseline | 0 | 1 | 0 | 3 | 2 | 2 | 4 | 6 | 0
  IgA ASC (aLT) - >2-fold increase over baseline | 2 | 5 | 5 | 5 | 4 | 6 | 7 | 10 | 6

3. Secondary Outcome: Antigen-Specific IgA Geometric Mean Titers
Description: Antigen-Specific IgA Geometric Mean Titers as defined by Fecal IgA. Final Clinical Study Report (FCSR) highlighted titer numbers only; no numbers for measure of dispersion/precision were given; no explanation as to why standard deviation information is not present in the FCSR.
Time Frame: Day 0, 21,42, 56, 70
Population: Only subjects receiving at least 2 vaccine doses were included in this assessment. Final Clinical Study Report (FCSR) highlighted titer numbers only; no numbers for measure of dispersion/precision were given; no explanation on not presenting standard deviation information is present in the FCSR.
Measure: Geometric Mean (Standard Deviation); unit: Geometric Mean Titers
Arm/Group | Group A-1 | Group A-2 | Group A-3 | Group B-1 | Group B-2 | Group C-1 | Group C-2 | Group D-1 | Group D-2
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 7 | 7 | 10 | 7
Geometric Mean Titers
  Day 0 - Anti-CfaE | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 9.56 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 43.66 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 11.34 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 21 - Anti-CfaE | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 8.77 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 5.94 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 9.63 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 59.75 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 16.95 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 42 - Anti-CfaE | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 12.06 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 22.99 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 162.67 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 56 - Anti-CfaE | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 44.22 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 4.29 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 52.52 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 23.47 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 70 - Anti-CfaE | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 9.47 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 8.63 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 18.12 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 8.98 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 190.44 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 0 - Anti-LT | 22.70 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 43.05 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 16.62 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 28.66 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 19.78 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 114.77 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 59.38 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 21 - Anti-LT | 15.00 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 189.39 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 13.89 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 46.07 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 19.82 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 9.85 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 16.56 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 137.37 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 51.60 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 42 - Anti-LT | 12.37 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 74.60 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 15.87 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 28.66 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 44.93 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 13.40 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 19.48 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 126.85 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 321.36 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 56 - Anti-LT | 33.30 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 83.68 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 18.16 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 31.53 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 40.24 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 23.00 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 23.35 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 142.69 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 27.83 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.
  Day 70 - Anti-LT | 13.15 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 98.89 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 9.54 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 7.59 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 31.27 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 17.38 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 82.77 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 266.20 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made. | 95.03 (NA) — The Final Clinical Study Report is the only record of available data, and no standard deviation data were included. Standard deviation data has not been located despite every effort made.

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group A-1 | Group A-2 | Group A-3 | Group B-1 | Group B-2 | Group C-1 | Group C-2 | Group D-1 | Group D-2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/7 | 0/7 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/7 | 0/7 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 5/5 | 5/5 | 7/7 | 7/7 | 10/10 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A-1 (N=5) | Group A-2 (N=5) | Group A-3 (N=5) | Group B-1 (N=5) | Group B-2 (N=5) | Group C-1 (N=7) | Group C-2 (N=7) | Group D-1 (N=10) | Group D-2 (N=8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related to vaccine
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Related to vaccine
GI symptoms (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Related to vaccine
Hemoglobin decrease (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Loose stools (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related to vaccine
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Right axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related to vaccine
Right knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Sleepiness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Tegaderm reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Related to vaccine
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to vaccine
Vaccine site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 5 (5) | 5 (5) | 1 (1) — Related to vaccine
Vaccine site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 5 (5) | 5 (5) | 6 (6) | 8 (8) | 8 (8) — Related to vaccine
Vaccine site reaction (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 5 (5) | 5 (5) | 5 (5) | 7 (7) | 7 (7) | 10 (10) | 8 (8) — Related to vaccine
Vaccine site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Related to vaccine
Vaccine site tenderness (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 6 (6) | 6 (6) | 8 (8) | 3 (3) — Related to vaccine
Vaccine site warmth (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Related to vaccine
Allergic rhinitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
ALT elevation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Ankle trauma, left (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
AST elevation (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to vaccine
Bilateral bicep strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
BP elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Creatinine elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Dorsal foot pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Unrelated to vaccine
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Generalized eruption, truncal proximal UE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 2 (2) — Unrelated to vaccine
Hemoglobin decrease (Investigations) | 0 (0) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 2 (2) — Unrelated to vaccine
Hemorrhoids (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Calf soreness, left (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Facial trauma, left eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Left metatarsal stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Left upper groin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) — Unrelated to vaccine
Menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Mental disorder NOS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Platelet decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccine
Ankel sprain, right (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Knee hyperflexion, right (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
RUE Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Scalp folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Allergies, seasonal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Unrelated to vaccine
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Subsurface blood clot, left calf (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to vaccine
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Tegaderm reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) — Unrelated to vaccine
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) — Unrelated to vaccine
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine
Viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to vaccine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No